CLINICAL TRIAL: NCT00294983
Title: OCD Among Patients With Burns
Status: Withdrawn | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Other Study IDs: SHEBA-05-3912-JZ-CTIL
Record Dates: First submitted 2006-02-19; First posted 2006-02-22 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Obsessive-Compulsive Disorder; Burns
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Burns

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Estimating the prevalence of OCD symptoms among patients with burns

ELIGIBILITY:
Inclusion Criteria:

* Patients with burns for at least 6 months and are under treatment

Exclusion Criteria:

* Was not defined

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Study Director — Sheba Medical Center; Nitsa Nacasch, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel